CLINICAL TRIAL: NCT03755622
Title: A Randomized Clinical Trial to Compare the Clinical Application of an Innovated Transpalatal Arch (TPA) Fabricated From 3D Reconstructed Model With Conventionally Constructed TPA.
Brief Title: Comparing Clinical Application of Innovatedly Made Transpalatal Arch (TPA) From 3D Reconstructed Model and Conventionally Made TPA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Wan Nurazreena Wan Hassan, Associate Professor, Lecturer at Department of Paediatric Dentistry and Orthodontics, Faculty of Dentistry, University of Malaya, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: DGD150005
Record Dates: First submitted 2018-10-30; First posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Transpalatal Arch (TPA); Oral Health Related Quality of Life (OHRQoL); Oral Health Impact Profile Short Version 14 (OHIP 14); Orthodontic Pain; Three Dimensional (3D) Orthodontic Device

STUDY DESIGN:
Intervention Model Description: Group C : Patients who receive Transpalatal Arch (TPA) that is conventionally constructed on stone models.
  Group 3D : Patients who receive Transpalatal Arch (TPA) fabricated from three dimensionally (3D) reconstructed study model.
Who Masked: Participant
Masking Description: Patients who received the Transpalatal Arch (TPA) are not aware whether the appliance is fabricated conventionally or made from 3D reconstructed study model.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C (Conventional) (Active Comparator): Group C consists of patients who receive Transplatal Arch (TPA) fabricated from conventionally made stone working model.
  Interventions: Device: Conventional Transpalatal Arch (TPA)
- Group 3D ( Three Dimensional) (Experimental): Group 3D consists of patients who receive Transpalatal Arch (TPA) made from 3D recontructed model.
  Interventions: Device: Transpalatal Arch (TPA) fabricated from 3D reconstructed model

INTERVENTIONS:
Device: Conventional Transpalatal Arch (TPA) — In Group C, upper molar bands selection will be carried out by direct intra oral procedure. The conventional TPA is made on the stone working models.
  Other Names: Conventionally made TPA
  Arms: Group C (Conventional)
Device: Transpalatal Arch (TPA) fabricated from 3D reconstructed model — In Group 3D, upper molar bands selection will be carried out on the 3D printed model instead of direct intra oral procedure. The 3D TPA will be fabricated on the 3D reconstructed model while the conventional TPA is made on the stone models.
  Other Names: TPA fabricated on 3D printed model
  Arms: Group 3D ( Three Dimensional)

SUMMARY:
Trans-palatal Arch or TPA is an intra oral device that is occasionally used in conjunction of orthodontic fixed appliance treatment. It has two main types, the fixed or removable TPA. The purpose of this appliance is to maintain upper jaw's arch width and preventing upper molar teeth from moving forward. It holds the upper molar teeth in their original position so that if any upper teeth are extracted to make room for the others to straighten, the upper molars will not move into the extraction spaces. It comprises of a stainless steel wire with a central semi loop that fits comfortably across but not touching the palate. On each side, it is attached with metal bands around each of the two upper molar teeth.

The construction of TPA requires at least three appointments that take up one to three weeks time. Firstly, an elastic "doughnut" like rubbery separators will be placed between the upper molar teeth using a special tool. Slight tightness is usually felt when the separators are inserted. The whole procedure takes less than a couple of minutes. Patients will be sent away for up to 14 days with the separators in place. For the second appointment, the separators will be removed with dental probe. The correct size metal bands are then selected for the upper molar teeth. Once a correctly fitting band has been chosen, an impression (mould) of the upper teeth with the bands in place will be taken. The impression, together with the bands will be sent to the laboratory for construction of the TPA. Separators will be placed again until patients come back to have TPA fitted.

If the mould of the teeth is scanned and printed out using three dimensions (3D) technology, the number of appointments could be reduced. The second appointment which requires molar bands selection, impression and replacement of separators of upper teeth could be skipped. Molar bands selection can be carried out outside the mouth and straight away sent to the laboratory for TPA construction. All parties involved, patients, clinicians and dental technologists will benefit the innovation by reduction of time spent for TPA related procedure. However, the study that compares innovated TPA from 3D reconstructed models and conventional method has never been done and related similar studies are very scarce.

DETAILED DESCRIPTION:
INTRODUCTION

Transpalatal Arch (TPA) has been invented by Dr. Robert Ara Goshgarian, a renowned orthodontist more than 7 decades ago. Throughout the years, various modifications of the design were made for different purposes and to increase its efficacy in achieving the optimum level of anchorage. In 1947, fabrication of Nance Palatal Ach (NPA) pioneered the adjustment of TPA by incorporation of an acrylic button that connects the palatal wire at the highest part of palatal vault. Recent innovations mostly involved adhesions of TPA to mini implants or temporary anchorage devices (TAD) and proven to be time and cost effective to be used in orthodontics. The usage of TPA for space maintenance demonstrated to be more advantagous in term of soft tissue compatibilty and increase in vertical control compared to Nance appliance. The combination of TPA and extraction of deciduos maxillary canines in the late mix dentition has shown to be an acceptable interceptive treatment to prevent maxillary canines palatal impaction. Despite numerous changes and alterations, the versatility of usage has made TPA remained as a useful adjunct in clinical orthodontics until today. However the fabrication of TPA required meticulous clinical steps which started with insertion of elastomeric separators on mesial and distal interproximal surfaces of maxillary permanent first molar teeth. One week later, separators were removed and series of molar bands selection or 'try in' session were carried out to get the correct size that fits the molar teeth. The drawbacks of this action is that, the 'used' molar bands if not properly decontaminated with an enzymatic cleaning and properly sterilized using autoclave, it may constitute a cross-infection hazard. An impression with molar bands in situ were taken and sent to the dental lab for fabrication of TPA followed by re-insertion of separators between the molar teeth. This means that each patient has to bear the discomfort caused by elastomeric separators for at least two weeks time or more. Orthodontists have to spent time for molar bands selection and dental technicians have more workload from pouring of impression until finishing of TPA.

RATIONALE

Patients do not have to undergo twice elastomeric separators placement as reported that among 4 orthodontic treatment procedures carried out,(upper alginate impression, separator placement, band placement and adjustment of arch wire), placement of separator causes a significant bacteraemia. Clinicians could cut down the number of appointments and time could be utilized to see more other cases. Currently there are 7 dental technicians in Paediatric and Orthodontic Department to cater for 10 Orthodontists, 6 Senior Postgraduates and 5 Junior Postgraduates, 1 technician was assigned for Optech management at Balai Ungku Aziz and starting from 2018, all technician will be involved in dental chair maintenance for the whole UM. Heavy workload and other commitments resulted in lack of time to finish all orthodontic cases.

AIM

To investigate whether TPA fabricated from 3D reconstructed model are feasible for clinical application.

OBJECTIVES

1. To compare the oral health related quality of life of patients before wearing TPA and after 3 months of appliance wear.
2. To compare the oral health related quality of life of patients wearing TPA fabricated from 3D reconstructed model and conventionally produced TPA up to 3 months.
3. To compare pain levels of patients wearing TPA fabricated from 3D reconstructed model and conventionally produced TPA up to 3 months.
4. To determine clinicians' preferences between TPA made from 3D reconstructed model and TPA produced from plaster dental cast.

PRIMARY OUTCOME

-Oral health related quality of life.

SECONDARY OUTCOME

* Pain levels.
* Clinicians preferences.

RESEARCH METHODOLOGY

Ethical Consideration:

* Ethical approval gained from Medical Ethics Committee, (DF CD1607/0057(P) Faculty of Dentistry, University of Malaya from 11th July 2016 - 31st May 2019
* Grant approved : PPPC/C1-2016/DGD/12 RM 17,085.00

Sample Size Calculation:

* Sample size estimation is based on comparative literature by (Johal et al., 2014) and calculated using G Power 3.1.92 software under supervision of statistician.
* Therefore, it was estimated that a sample size of 46 subjects was needed to demonstrate a significant change in OHRQoL, with an 80 per cent probability power at the 5% level of significance.
* The sample size was inflated by a 10% margin to allow for loss to follow-up and drop outs; thus, the total sample size was a minimum of 52.

MATERIAL AND METHODS

52 patients undergoing orthodontic treatment at Orthodontic Clinic, University of Malaya, required Transpalatal Arch (TPA) and fulfilled the inclusion criterias will be be randomly selected for this single-blinded study.They will be divided into two groups (n =26 for each group) , Group C will received conventional TPA while Group 3D will be given TPA fabricated on three-dimensionally (3D) reconstructed model. 6 orthodontic postgraduates will be involved in providing treatment for these patients. 4 operators will be having 9 patients each while the other 2 operators will have 8 patients each. 4 operators will be provided with an opaque envelope comprises of 9 lots each and 2 operators will have 8 lots each. Dental Surgery Assistant (DSA) assisting each operator will open the opaque envelope that have been allocated for each sample after the written consent is signed.Baseline questionnare (T0) will be distributed at this stage, prior to fabrication of TPA. Group C will undergo normal clinical and laboratory procedure of conventional TPA. For Group 3D, the dental casts will be sent to Centre For Biomedical And Technology Integration (CBMTI) for digitization using the Geomagic Capture three-dimensional scanner carried out by 2 trained Design Engineer.Captured images are automatically processed by the Geomagic Design X software and virtually remodelled by the same personnel. Total resection of upper right and left second premolars (15, 25) and upper right and left second molars (17, 27) were simulated prior to printing for easier molar band insertion and cost reduction. Modified 3D dental model were printed out using Acrylonitrile-Butadine-Styrene (ABS) material through Fused Deposition Modelling (FDM) technique . TPA will be constructed on it by the same technician who fabricated the conventional version. First modified OHIP 14, (T1) will be distributed 1 week post cementation of TPA, followed by T2 at 1 month post insertion and T3 at 3 months post cementation. Patients will be dismissed from the study after the T3 stage.

SELECTION CRITERIA

Patients requiring TPA in conjunction with upper and lower FA

CONSENT All patients were given oral and written information concerning the study and signed a written consent

INCLUSION CRITERIA

* Age 18 and above
* Requiring premolar extractions
* Patients do not have previous orthodontic treatment before

EXCLUSION CRITERIA

* Patient requiring lingual arch, modified TPA, Nance Palatal Arc
* Non extraction upper arch treatment
* Patients requiring upper arch expansion
* Requiring upper first permanent molar extraction
* Presence of dento-facial anomalies.
* Patients requiring orthognathic surgery

MEASURING METHODS AND DATA COLLECTION

Acquisition of digital model:

-Conventional study model will be scanned using structured light scanner (Geomagic Capture) to produce 3D digital model.

Virtual remodelling :

-Simulated cutting of upper second premolar and upper second molar teeth via Geomagic Design X (XOR) software prior to printing to reduce the cost.

Printing of 3D reconstructed model :

A 3D "UP Plus 2" printer will print out the remodeled version with Acrylonitrile Butadiene Styrene (ABS) material.

Construction of TPA :

All TPAs will be constructed by the same technician, using the same type of Molar Bands (3M Unitek), 0.9 stainless steel wire and similar type of cementation that is 3M Unitek Multi-Cure Glass Ionomer Orthodontic Band Cement.

Randomization

https://www.randomizer.org/

Measuring tools

* OHIP Questionnaires adapted from: Oral Health Impact Profile Malaysian version (S-OHIP[M]).
* The respondents are asked to answer on a five-point frequency Likert scale (very often, quite often, sometimes, once a while, and never).
* Progress record of each device to operators.
* Focus group discussion (FGD) among 5 operators.

Statistical Analysis

* Statistical Package for Social sciences (SPSS version 22.0.0.0)
* Analysis : Paired t-test, Repeated measure ANOVA
* Qualitative analysis : NVivo

OHIP

* Oral Health Impact Profile Malaysian version (L-OHIP[M]) with 45 items is an adaptation of the original version developed by Slade and Spencer (1994), 49 items
* Short version (S-OHIP[M]) was also developed, which contains only 14 items -Seven domains namely:-

  1. Functional limitation
  2. Physical pain
  3. Psychological discomfort
  4. Physical disability
  5. Psychological disability
  6. Social disability
  7. Handicap

Although the S-OHIP(M)was developed to be used as a descriptive and discriminative measure in population oral health surveys, it may also be appropriate for use in clinical trials and in clinical practice as an evaluative measure.

FOCUS GROUP DISCUSSION

* Focus group interview is a "carefully planned discussion designed to obtain perceptions in a defined area of interest in a permissive, nonthreatening environment" (Krueger, 1988).
* Intended to promote self disclosure among participants.
* Most likely to happen when the participants perceive that they are alike in some important way and when the environment is non judgmental.
* 6 - 10 participants, 1 moderator.
* Conversation taped, recorded.
* 60 - 90 minutes.
* Until saturation point reached (saturation is the point at which no new information emerges).
* Transcribe into several themes.
* Analyze by NVivo software.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and above
2. Requiring premolar extractions
3. Patients do not have previous orthodontic treatment before

Exclusion Criteria:

1. Patient requiring lingual arch, modified TPA, Nance Palatal ArchNon extraction upper arch treatment
2. Patients requiring upper arch expansion
3. Requiring upper first permanent molar extraction
4. Presence of dento-facial anomalies.
5. Patients requiring orthognathic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2017-06-11 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Change of oral health related quality of life between patients wearing conventional TPA and TPA fabricated from 3D reconstructed model from baseline and at 3 months of wear. | 3 months
  To compare the level of Oral health related quality of life (OHRQoL) between patients wearing conventional Transpalatal Arch and patients wearing Transpalatal Arch fabricated from three dimensionally reconstructed model in three interval times that is after 1 week (T1) , 1 month (T2) and up to three months post Transpalatal Arch cementation (T3). This is achieved by using validated short version Oral Health Impact Factor 14 (OHIP) questionnaire as the instrument. The minimum score per indivudual is 14 and the maximum score is 70. The lesser the score, the better oral health realted quality of life the patient has.

SECONDARY OUTCOMES:
Change of pain level from baseline to 3 months of wear between patients wearing conventional TPA and TPA fabricated from 3D reconstructed model. | 3 months
  Pain levels between patients in the two groups, Group C (Conventional) and Group 3D (TPA on fabricated from three dimensionallay recontructed model) is compared using quesitionnaire with visual analog score (VAS) and Likert Scale at 1 week (T1), 1 month (T2) and three months (T3) post insertion of the Transpalatal Arch. Score 0 indicating no pain, score 1 to 3 indicating mild pain , score 4 to 6 showing moderate level of pain and score 7 to 9 for severe pain. The minimum score is zero and maximun score is 10. The higher the score, the higher the pain level is.
Qualitative evaluation of clinicians preferences regarding clinical application between the conventional TPA and TPA fabricated from 3D reconsructed model. | 3 months
  Six clinicians (who delivered the device to both group of patients) preferences' between the conventional Tranpalatal Arch and Transpalatal Arch made from three dimensionally reconstructed model is assessed through focus group discussion (FGD). The FGD will be conducted by one moderator with presence of a transcriber. The discussion will end after the point of saturation is met, that is the point where there is no more new issues brought up by the clinicians. The whole discussion will be recorded and transcribed by the third party and content will be analyzed in qualitative manner.

CONTACTS AND LOCATIONS:
Locations (1):
- Postgraduate Orthodontic Clinic, Faculty of Dentistry, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No